CLINICAL TRIAL: NCT05763485
Title: Anti Reflux Mucosal Ablation Therapy in PPI Dependent GERD: a Prospective Randomized, Single-blinded, Sham-controlled Trial
Brief Title: Anti Reflux Mucosal Ablation Therapy in PPI Dependent GERD
Acronym: APDG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Mohamed Abdelhafez, Principal Investigator Dr. Abdelhafez, Technical University of Munich
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R0001
Record Dates: First submitted 2023-02-09; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Gastroesophageal Reflux
Keywords: anti reflux mucosal ablation; ARMA
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: 4 months after the initial procedure (ARMA or sham-procedure) patients are unblinded. Patients who initially received the sham procedure are now allowed to be treated by ARMA.
Who Masked: Participant
Masking Description: Patients are randomized equally into an intervention and control group. The patients remain blinded to the procedure until 4 months after the initial procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti reflux mucosal ablation (ARMA) (Active Comparator): Patients randomized into the intervention arm receive ARMA and a follow up control after 2, 4, 6 and 12 months. PPI treatment is stopped after 2 months until the end of the study or worsening of symptoms. Esophagogastroduodenoscopy, manometry and pH metry is performed after 4 months.
  Interventions: Procedure: Anti reflux mucosal ablation (ARMA)
- Sham procedure (Sham Comparator): Patients randomized into the sham procedure arm receive a esophagogastroduodenoscopy in the same setting as if ARMA would be performed. Patients in the Control group receive follow up controls after 2 and 4 months and after unblinding after 4 months are allowed to perform a crossover to receive ARMA. PPI treatment is stopped 2 months after the initial sham procedure until the end of the study or worsening of symptoms. If the patients receive ARMA as a crossover reevaluation is performed 2, 4, 6 and 12 months after the actual ARMA procedure.
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Anti reflux mucosal ablation (ARMA) — In patients fulfilling the inclusion criteria and being randomized for ARMA, the procedure using argon plasma coagulation involves two semicircular ablations of the mucosa of the EGJ in a butterfly shape of a width of 2 cm. The approximate duration of the procedure is 30min.
  Follow includes objective evaluation of reflux disease by reflux questionnaires, esophagogastroduodenoscopy, esophageal manometry, pH metry.
  Arms: Anti reflux mucosal ablation (ARMA)
Procedure: Sham procedure — In patients fulfilling the inclusion criteria and being randomized for sham procedure, the procedure involves esophagogastroduodenoscopy with the same set of movements and duration as the ARMA procedure without the actual ablation.
  Arms: Sham procedure

SUMMARY:
This is a prospective, randomized, single-blinded, interventional, controlled trial to evaluate the efficacy and safety of endoscopic anti reflux mucosal ablation (ARMA) in PPI dependent gastroesophageal reflux disease (GERD) in comparison to controls with a sham procedure.

DETAILED DESCRIPTION:
Patients who fulfill the inclusion criteria and, after informed consent, are willing to participate in this study will be prepared for ARMA. After sedation the patients will be randomized equally into an intervention and control Group. The patients are blinded to the procedure. The Patients in the intervention group receive ARMA using argon plasma coagulation (APC) at the gastroesophageal junction (EGJ) in two semicircular patterns while the control group receives a sham procedure. The approximate duration of the procedure is 30min. After the procedure the patients receive follow up controls at 2, 4, 6 and 12 months. During the first follow up, 2 months after the procedure symptoms are evaluated by questionnaires (GERD- HRQL, FSSG, VAG). Subsequently the PPI- medication is stopped in all patients until the end of the study or worsening of symptoms. During the second follow up 4 months after the initial procedure the symptoms are reevaluated by questionnaires. The patients are then unblinded and are told if they received ARMA or sham procedure. Those patients who received ARMA are examined by esophagogastroduodenoscopy, esophageal manometry and pH metry. Further assessments is performed by questionnaires 6 and 12 months after the initial procedure.

Those patients in the control group are allowed to take part in a crossover to receive the ARMA procedure as well. If they receive ARMA, symptoms are reevaluated 2 months after the procedure by questionnaires, esophagogastroduodenoscopy, esophageal manometry and pH metry. Further controls are performed after 4, 6 and 12 months by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* PPI dependent GERD for at least 6 months
* Pathological esophageal acid exposure, defined by DeMeester score >14.7 or acid exposure time (AET) >4.2% in pH metry while off PPI
* Exclusion of primary esophageal motility disorders by manometry
* Upper endoscopy with biopsy (Exclusion of eosinophilic esophagitis)

Exclusion Criteria:

* Sliding hiatal hernia >3cm
* Los Angeles grade C/D esophagitis
* Primary esophageal motility disorders
* Grade IV Hill´s flap valve
* Pregnancy or planed pregnancy in the next 12 months
* Eosinophilic esophagitis
* Paraesophageal hernia
* Previous esophageal or gastric surgery
* Barretts esophagus
* Liver cirrhosis
* Varices
* Lack of consent
* ASA physical status >III

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in symptoms of gastro esophageal reflux disease | 4 months
  Improvement in symptoms of gastro esophageal reflux disease by more than 50% from baseline in GERD-Health Related Quality of Life Questionnaire (GERD- HRQL) at 4 months after procedure. Total score 0-50; higher scores indicate greater complaints.

SECONDARY OUTCOMES:
Change in symptoms of gastro esophageal reflux disease | 12 months
  Change in symptoms of gastro esophageal reflux disease in GERD-Health Related Quality of Life Questionnaire (GERD- HRQL) at 6 and 12 months. Total score 0-50; higher scores indicate greater complaints.
Change in symptoms of gastro esophageal reflux disease | 12 months
  Change in symptoms of gastro esophageal reflux disease in regurgitation score at 4, 6 and 12 months. Total score 0-30; higher scores indicate greater complaints.
Change in symptoms of gastro esophageal reflux disease | 12 months
  Change in symptoms of gastro esophageal reflux disease in Frequency scale for the symptoms of GERD (FSSG) at 4, 6 and 12 months. Total score 0-48; higher scores indicate greater complaints.
Change in symptoms of gastro esophageal reflux disease | 12 months
  Change in symptoms of gastro esophageal reflux disease in visual analog scale (VAS) at 4, 6 and 12 months. Total score 0-10; higher scores indicate greater complaints.
Complication rate | 12 months
  Recording of all complications in relation to the ARMA- procedure
PPI dependency | 12 months
  Requirement and dose of PPI at 4, 6 and 12 months
Change in esophageal acid exposure at 4 months after ARMA | 4 months after ARMA
  Change in esophageal acid exposure in pH metry 4 months after ARMA
Change in lower esophageal sphincter pressure 4 months after ARMA | 4 months after ARMA
  Change in lower esophageal sphincter pressure in manometry 4 months after ARMA
Postinterventional pain | 1day
  Recording of postinterventional pain in visual analog scale (VAS). Higher scores indicate greater complaints.
Changes in cardia morphology | 4 months after ARMA
  Changes in Hill's flap grade
Technical success rate | 1 day
  Successful completion of ARMA

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelhafez, MD, Principal Investigator — Universitiy Hospital Rechts der Isar, Technical Universitiy Munich
Locations (1):
- II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No